CLINICAL TRIAL: NCT02494128
Title: Early Group Based Parental Support Within Child Health Service - Group Leadership
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skåne, Centre of Excellence for Child health care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H152014/397
Record Dates: First submitted 2015-05-04; First posted 2015-07-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Family Health
Keywords: Child health service; Family health; Nurse; Education; Parental group; Group leadership; Health promotion
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Education in group leadership
  Interventions: Other: Education
- Control group (No Intervention): This group fills in the questionnaire. No intervention given.

INTERVENTIONS:
Other: Education — Education in group leadership
  Arms: Intervention group

SUMMARY:
All parents in Sweden are offered group based parental support within Child Health Service (CHS) but only 40% participate. Nurses feel insecure in their group leadership and express a need for education in group leadership and group dynamics. Most CHC nurses do not have formal education or training in group leadership and the aim of this study was to evaluate a group based education program in group leadership for Child Health Care (CHC) nurses.

DETAILED DESCRIPTION:
The study follows the guidelines for complex interventions (MRC) and was set up as a randomized controlled trial (RCT) evaluated with questionnaires before and after the intervention. Focus group interviews 6 months after the intervention will be performed with the CHC nurses participating in intervention group. 3 groups with 25 CHC nurses in each group are to participate in a three day education in group leadership and group processes. The education aims to provide knowledge and awareness about group dynamics, group processes and group leadership and also aims towards increased self-awareness in the role as group leader.

ELIGIBILITY:
Inclusion Criteria:

* working within child health service in Skåne, Sweden
* managing at least 2 parental groups/year

Exclusion Criteria:

* no parental groups

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in experience of group leadership | 2 weeks before and 6 months after the education
  Change in experience of group leadership will be measured by a previously used questionnaire (Wallby, T (2008) parental support un Sweden today - What, when and how. Swedish National Institute of Public Health. (Föräldrastöd i Sverige idag - Vad när hur?) and Lefevre et al, 2013. Managing parental groups during early childhood: New challenges faced by Swedish child health nurses. Journal of child health care).The questionnaire consists of 38 questions concerning structure, content and extent of parental groups as well as questions about group leadership and background characteristics. Analysis will be performed using Statistical Package for Social Sciences (SPSS) and will be presented in a descriptive way
Relevance and experience of the education in group leadership | After completed intervention, intervention has an expected average duration of 12 weeks.
  A course evaluation form previously used in educations with primary health care nurses will be completed after the intervention is completed, before leaving site. It consists of seven questions about the content and relevance of the course.Four questions were arranged with a 5-point Likert scale ranging from 1 "poor" to 5 "excellent", and three questions were open-ended given the possibility to respond in free text.The numeric questions will be summarised and presented descriptive and the answers in text will be analysed by content analysis in a manifest way.
Change in experience of group leadership and relevance and experience of the education in group leadership | 6 months after the education
  Change in experience of group leadership and relevance and experience of the education in group leadership will be explored in Focus group interviews with at least 3 focus groups. The interviews will be analysed by manifest and latent content analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hallström, Professor, Principal Investigator — Child, family and reproductive health, University Lund

IPD SHARING:
Plan to Share IPD: Yes
Two articles will be published presenting the results.

REFERENCES:
- [Derived] Silva JAM, Mininel VA, Fernandes Agreli H, Peduzzi M, Harrison R, Xyrichis A. Collective leadership to improve professional practice, healthcare outcomes and staff well-being. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD013850. doi: 10.1002/14651858.CD013850.pub2. PMID 36214207
- [Derived] Lefevre A, Lundqvist P, Drevenhorn E, Hallstrom I. "From resistance to challenge": child health service nurses experiences of how a course in group leadership affected their management of parental groups. BMC Nurs. 2017 Dec 2;16:73. doi: 10.1186/s12912-017-0267-6. eCollection 2017. PMID 29213213